CLINICAL TRIAL: NCT01215487
Title: A Study Investigating the Predictive Value of Philadelphia Positive Stem Cell Properties in Newly Diagnosed Patients With Chronic Myeloid in Chronic Phase Receiving Treatment With Imatinib
Brief Title: A Study Investigating the Predictive Value of Philadelphia Positive Stem Cell Properties in Newly Diagnosed Patients With Chronic Myeloid Leukemia in Chronic Phase Receiving Treatment With Imatinib
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Donna Forrest, Principal Investigator, University of British Columbia
Other Study IDs: H09-03255
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML Predictive Study
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens of whole blood will be collected, and used for measurement of sensitivity of the patient's individual pretreatment colony-forming cells (CFCs) to IM exposure in vitro, the level of expression of BCR-ABL, OCT1, ABCB1/MDR and ABCG2 transcripts in their CD34+ cells and the frequency of mutant BCR-ABL transcripts in the same cells. The cells are cultured for 3 weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 - Chronic Myelogenous Leukemia Patients: Patients will be selected from patients referred to the primary hospital site for treatment and assessment. The patients will be approached by the physicians and or the study research nurse to consider participation in the study. Patients may be selected by participating off-site hospital centres and may be enrolled at those collaborating centres.
  Interventions: Procedure: Stem Cell and Mutational Assay

INTERVENTIONS:
Procedure: Stem Cell and Mutational Assay — Laboratory blood testing

SUMMARY:
Imatinib (IM) is first-line treatment for patients with newly diagnosed CML in chronic phase. The drug is associated with high rates of cytogenetic responses with minimal toxicity in approximately 80% of patients. In 20% of patients however, the disease is either initially unresponsive to IM (Imatinib), resistance develops within a few months, or blast crisis occurs early and unexpectedly following an initial response. An increasing body of clinical evidence indicates that single agent molecularly targeted therapy (as in Gleevec/Imatinib) will not cure most patients with CML, as molecular remissions are rare. There is currently no clinically useful predictive tests to identify AT DIAGNOSIS those patients who are destined to be IM failures. The authors of this study have recently demonstrated that CML stem/progenitor cells are biologically insensitive to IM and are also genetically unstable and rapidly generate IM-resistant mutants in vitro and in vivo. The team recently discovered that the CD34 stem/progenitor cells of newly diagnosed CML patients who subsequently fail to respond to IM treatment show a reduced response to IM and a higher frequency of BCR-ABL mutations by comparison of 14 IM non-responders with 11 IM-responders. If this finding can be validated in a larger prospective cohort of patients, this predictive test could be used to more rationally design treatment plans with early addition of alternative therapies ie: Dasatinib or combination therapies for patients according to their individual risk profiles.

Hypothesis:

The clinical response of newly diagnosed chronic phase CML patients to IM can be predicted by certain biological properties of their CD34 stem/progenitor cells which are variable among patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CML in chronic phase.
* ECOG <2.
* Normal organ function and ULN Total bili, AST and ALT.
* Must have the ability to understand and sign a written consent form

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* May not have prior treatment with Imatinib, Dasatinib, Nilotinib or other tyrosine kinase inhibitors.
* Patients must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing mothers
* Patients must have no prior malignancies except for; adequately treated non-melanoma skin cancer, cervical carcinoma-in-situ, adequately treated Stage I or II cancer from which the patient is in complete remission, or any other cancer from which the patient has been disease free for 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from patients referred to the primary hospital site for treatment and assessment. The patients will be approached by the physicians and or the study research nurse to consider participation in the study. Patients may be selected by participating off-site hospital centres and may be enrolled at those collaborating centres.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-10; Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Jiang, Study Director — University of British Columbia - Terry Fox Laboratory; Ryan Brinkman, Study Director — University of British Columbia - Terry Fox Laboratory; Connie Eaves, Study Director — University of British Columbia - Terry Fox Laboratory; Lynda Foltz, Study Director — University of British Columbia - St. Paul's Hospital Department of Hematology
Locations (1):
- Leukemia BMT program of BC, Vancouver General Hospital, Hematology Research and Clinical Trials Unit, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Related Info — http://www.leukemiabmtprogram.com